| Examination of the Effects of Chromium Levels on Glucose Metabolism, Lipid |
|-----------------------------------------------------------------------------|
| Metabolism, Morbidity and Mortality Rates in Patients Followed in Intensive |
| Care Unit |

Hacettepe University, Department of Anesthesiology and Intensive Care

Turkey

ClinicalTrials.gov #NCT06334042

Document Date: 24 December 2024

This study was approved by the Hacettepe University Non – Interventional Clinical Research Ethics Committee on July 25, 2023, with the reference number GO 23/488 (Decision Number: 2023/13 – 54) and was supported by the Hacettepe University Scientific Research Projects Coordination Unit (Project Number: 21026). The study is non – interventional, prospective, and observational. It included 309 patients followed in the Anesthesiology Intensive Care Unit of Hacettepe University Hospital between February 7, 2024, and August 8, 2024.

## **Study Location**

The evaluation of patients for eligibility, recording of parameters, and collection of blood samples were conducted in the Anesthesiology Intensive Care Unit of Hacettepe University Hospital.

Lipid profile and HbA1c measurements were performed in the Department of Biochemistry Laboratory of the same hospital. Blood samples for chromium measurement were also stored in this laboratory before analysis.

Blood chromium levels were measured at the Department of Pharmaceutical Toxicology, School of Pharmacy, Hacettepe University.

## Study Population, Sample, and Research Group

#### **Inclusion Criteria**

- Age ≥ 18 years,
- Being followed up in the Anesthesiology Intensive Care Unit of Hacettepe University Hospital,
- Availability of required data (medical history, laboratory results, etc.) for analysis,
- Not taking chromium supplements.

#### **Exclusion Criteria**

- Age < 18 years,</li>
- Refusal to participate in the study,
- Taking chromium supplements.

### **Research Method and Data Collection Tools**

Data of patients meeting the inclusion criteria in the Anesthesiology Intensive Care Unit were obtained from: blood samples sent to the laboratory during the patient's stay, medical history collected from the patient or relatives, and nurse follow – up forms. The patients were followed up by Dr. Oğuzhan KAHVECİ during their stay, with data recorded both physically and digitally. Blood samples were sent to the laboratory weekly, starting from the patient's admission.

### **Data Collection**

### **Data Collection**

Parameters shown in Table 1 were monitored throughout the ICU stay.

## **Table 1. Data Collection Form**

| Parameters | Timing |
|--------------------------|---------------------------|
| Date | Upon Admission and Weekly |
| Age | Upon Admission |
| Gender | Upon Admission |
| Height (cm) | Upon Admission |
| Weight (kg) | Upon Admission |
| Body Mass Index (BMI) | Upon Admission |
| Comorbidities | Upon Admission |
| Reason for ICU Admission | Upon Admission |
| SOFA Score | 24 Hours Post-Admission |
| APACHE – II Score | Upon Admission |
| Nutritional Status | During Stay |
| Triglycerides (mg/dL) | Upon Admission and Weekly |

Parameters Timing

HDL (mg/dL) Upon Admission and Weekly

LDL (mg/dL) Upon Admission and Weekly

VLDL (mg/dL) Upon Admission and Weekly

Total Cholesterol (mg/dL)

Upon Admission and Weekly

HbA1c (%) Upon Admission

Blood Glucose (mg/dL)

Daily During Stay

Coefficient of Variation (CV) (%)

During Stay

Blood Chromium Level (µg/L)

Upon Admission and Weekly

ICU Stay Duration Throughout ICU Stay

Post-Discharge Outcome (Discharge, Transfer, Death) Upon Discharge

Hospital Stay Duration ICU and Ward Duration

## **Power Analysis**

Based on a study by Chen et al., which examined plasma chromium levels in relation to metabolic syndrome components in a large patient group, the effect size (Cohen's D) was calculated as 0.202. With a 0.05 error margin and 0.95 power, the minimum sample size required to detect significant differences in repeated measures was calculated as 277. The sample size estimation was performed using G\*Power 3.1.9.7.

# **Blood Sample Analysis**

## **Capillary Blood Glucose**

Measurements (mg/dL) taken from fingertip blood by nurses using FreeStyle Optium Neo H glucometer and Abbott Blood Glucose Test Strips.

## **Lipid Profile**

Triglycerides (mg/dL), Total Cholesterol (mg/dL), HDL (mg/dL), LDL (mg/dL), and VLDL (mg/dL) were analyzed in the Beckman Coulter AU 5800 device in the Biochemistry Laboratory.

### HbA1c

Analyzed (%) using the Tosoh G11 device in the Biochemistry Laboratory.

### **Blood Chromium Level**

Analyzed (µg/L) using the Thermo Scientific iCAP Q ICP – MS device in the Department of Pharmaceutical Toxicology, School of Pharmacy.

# **Statistical Analysis**

Data were analyzed using IBM SPSS Statistics 25 © Copyright SPSS Inc. 1989, 2017. Normal distribution of continuous variables was examined using Kolmogorov – Smirnov and Shapiro – Wilk tests, depending on sample size. Categorical variables were presented as frequency (n) and percentage (%), and continuous variables were expressed as mean ± standard deviation (SD), median (IQR 25 – 75), and minimum – maximum values. Mann – Whitney U test, a non – parametric test, was used for analyzing independent two – group data as the data did not show normal distribution. Pearson Chi – Square Test, Fisher's Exact Test, Fisher's Freeman – Halton Exact Test, Yates' Correction, and Post – Hoc Bonferroni adjustments were used for independent categorical variable analysis. For correlation analysis between continuous variables, Spearman Rho Correlation Analysis was applied. Friedman Test and Post – Hoc Bonferroni adjustments were used for comparing dependent variables in more than two groups when parametric test assumptions were not met. Statistical significance was set at 0.05.